CLINICAL TRIAL: NCT05964556
Title: The Relationship Between The Functional Movement Screen and Isokinetic Muscle Strength of Knee in Different Sport Branches
Brief Title: Relationship Between the Functional Movement Screen and Isokinetic Muscle Strength of Knee in Different Sport Branches
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, TUĞBA BİRBEN, research assistant, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2017/23
Record Dates: First submitted 2023-07-16; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Muscle Strength; Sport Injury; Muscle Contraction
Keywords: Functional movement screen; H/Q ratio; isokinetic systems; muscle strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Functional Movement Screen and Isokinetic Muscle Evulation of Knee Muscles: Functional movement screen was evaluated with 7 basic parameters determined by Gray Cook Isokinetic muscle measurements were performed with an ISOMED 2000
  Interventions: Other: Functional Movement Screen (FMS); Other: Isokinetic Muscle Evulation of Knee Muscles

INTERVENTIONS:
Other: Functional Movement Screen (FMS) — FMS is an analysis system that evaluates muscle strength imbalance and functional performances on the dominant-non-dominant side in athletes. It aims to detect stability and mobility that can be ignored in the asymptomatic active population and athletes. It consists of 7 basic parameters determined by Gray Cook (Deep Squat, Hurdle Step, -In-line Lunge, Shoulder Mobility, Active Straight Leg Raise, Trunk Stability, Rotatory Stability). The athletes were evaluated after giving verbal instructions to the athletes about the head, trunk, knee and foot positions. For each parameter, the athletes were given points between 0-3 values. The total score was determined as 21 points. Completing the movement completely and without compensation was given 3 points, and 2 or 1 points were given according to the activation of the compensation mechanism and balance disorders. In case of any pain during or at the end of the movement in the evaluated parameter, 0 points were given to the athletes.
Other: Isokinetic Muscle Evulation of Knee Muscles — The isokinetic knee flexor and extensor group muscle strengths of the athletes participating in the study were measured on the dominant and non-dominant sides. Measurements were performed with an ISOMED 2000 (D&R Ferstl GmbH, Hemau, Germany) isokinetic measuring device. The test protocol was adjusted to be concentric/concentric. Measurements were made at angular velocities of 60°/sec and 180°/sec. At an angular speed of 60°/sec, the athlete was asked to perform 10 repetitions of voluntary knee flexion/extension at maximum strength. Then, after resting for 30 seconds, 30 repetitions of knee flexion/extension were performed at an angular velocity of 180°/sec. Before starting the test in both angular speeds, 3 repetitive attempts were made to learn the movement. The following parameters were evaluated at 60°/sec and 180°/sec angular speed.

SUMMARY:
This study was conducted to demonstrate the correlation between the functional movement screen and the isokinetic muscle strength with objective data. Investigators conclude that the use of FMS in combination with isokinetic systems will provide more detailed information on the prevention of injuries to sports and the improvement of performance.

DETAILED DESCRIPTION:
This study was conducted to demonstrate the correlation between the functional movement screen and the isokinetic muscle strength with objective data. 60 athletes involved in volleyball, greco-roman, speed skating, athletics and taekwondo branches were included in the study. The functional movement of the athletes was assessed by Functional Movement Screening, lower extremity isokinetic muscle strength was assessed by ISOMED 2000® isokinetic device.

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily agreed to participate in the study
* Have at least 3 years of licensed sports experience

Exclusion Criteria:

* Those who have had or have ongoing orthopedic problems in the last 6 months

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Carried out with 60 athletes between the ages of 12-30 who are interested in different or same sports branches.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Funtional Movement Screen (FMS) | 20 minutes
  FMS is an analysis system that evaluates muscle strength imbalance and functional performances on the dominant-non-dominant side in athletes. It aims to detect stability and mobility that can be ignored in the asymptomatic active population and athletes. It consists of 7 basic parameters determined by Gray Cook (Deep Squat, Hurdle Step, -In-line Lunge, Shoulder Mobility, Active Straight Leg Raise, Trunk Stability, Rotatory Stability). The athletes were evaluated after giving verbal instructions to the athletes about the head, trunk, knee and foot positions. For each parameter, the athletes were given points between 0-3 values. The total score was determined as 21 points. Completing the movement completely and without compensation was given 3 points, and 2 or 1 points were given according to the activation of the compensation mechanism and balance disorders. In case of any pain during or at the end of the movement in the evaluated parameter, 0 points were given to the athletes.
Isokinetic Measurement of Knee Muscles | 20 minutes
  The isokinetic knee flexor and extensor group muscle strengths of the athletes participating in the study were measured on the dominant and non-dominant sides. Measurements were performed with an ISOMED 2000 (D&R Ferstl GmbH, Hemau, Germany) isokinetic measuring device. The test protocol was adjusted to be concentric/concentric. Measurements were made at angular velocities of 60°/sec and 180°/sec. At an angular speed of 60°/sec, the athlete was asked to perform 10 repetitions of voluntary knee flexion/extension at maximum strength. Then, after resting for 30 seconds, 30 repetitions of knee flexion/extension were performed at an angular velocity of 180°/sec. Before starting the test in both angular speeds, 3 repetitive attempts were made to learn the movement. The following parameters were evaluated at 60°/sec and 180°/sec angular speed.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA BIRBEN, PhD, Study Director — Recep Tayyıp Erdogan University Guneysu Vocational School of Physical Therapy and Rehabilitation
Locations (1):
- Recep Tayyıp Erdogan University Guneysu Vocational School of Physical Therapy and Rehabilitation, Rize, Guneysu, Turkey (Türkiye)